CLINICAL TRIAL: NCT00644202
Title: A Pilot Weight Control Intervention at Harvard Pilgrim Health Care (HPHC)
Brief Title: A Pilot Weight Control Intervention at HPHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Harvard Pilgrim Health Care (Other)
Responsible Party: Gary Bennett, Ph.D, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-007
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Obesity
Keywords: weight control
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Intervention Group
  Interventions: Behavioral: Counseling Sessions; Behavioral: Specialized Website; Behavioral: Telephone Counseling Calls
- Group 2 (No Intervention): Usual Care Group

INTERVENTIONS:
Behavioral: Counseling Sessions — Counseling Sessions at each study visit around diet and physical activity from a registered dietician
  Arms: Group 1
Behavioral: Specialized Website — Specialized website that allows participants to track their eating and physical activity patterns, learn new weight management skills, interact with the dietician, and receive support from other participants
  Arms: Group 1
Behavioral: Telephone Counseling Calls — 5 telephone calls with a health counselor, lasting 15-20 minutes each.
  Arms: Group 1

SUMMARY:
The purpose of this study is to examine how adults can improve their physical activity levels and eating habits using an interactive web-based weight control program and regular contact with a dietician.

DETAILED DESCRIPTION:
* All study participants must have regular access to the Internet, however, the study will not provide this access. Participants will be randomly placed in one of two study groups (Group 1 or Group 2).
* Group 1 participants will be asked to make 3 in-person visits, each lasting 75-90 minutes. The following information will be collected: name, mailing address, telephone number, and email address. During the study visit, the following measurements will be taken: height, weight, waist circumference, blood pressure and dietary patterns.
* Group 1 participants will also receive counseling around diet and physical activity from a registered dietician and be asked to use a specialized website that will allow them to track eating and physical activity patterns, learn new weight management skills, interact with the dietician, and receive support from other participants.
* Group 1 will also receive 5 telephone counseling calls with a health counselor. During the telephone calls, we will teach the participant new skills such as tracking diet and physical activity, goal-setting and staying motivated.
* Group 2 participants will be asked to make 2 in-person visits, each lasting 75-90 minutes in length. The following information will be collected: your name, mailing address, and telephone number. During the study visit, the following measurements will be taken: height, weight, waist circumference, blood pressure and dietary patterns.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 65 years of age
* Body mass index between 30-40 kg/m2
* Non-smoker (quit within previous 6 months)
* Comfort reading and speaking English
* Stage 1 hypertension
* Not currently pregnant
* Regular web access from home

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Weight | 24 weeks

SECONDARY OUTCOMES:
Blood pressure | 24 weeks
Diet | 24 weeks
Physical activity | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bennett, Ph.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Department of Ambulatory Care and Prevention, Boston, Massachusetts